CLINICAL TRIAL: NCT06378567
Title: A Between Groups, Placebo-controlled US Home Placement Study Designed to Assess the Effects of Dietary Supplement Drinks on Sleep, Stress and Mood
Brief Title: A Study to Assess the Effects of Dietary Supplement Drinks on Sleep, Stress and Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Water Street Collective (Industry)
Collaborators: British American Tobacco (Investments) Limited (Industry); HCD Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HCD J8923
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-08

CONDITIONS: Sleep; Mood; Stress

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo comparator (Placebo Comparator): Investigational liquid shot beverage product: prototype 60ml product that does not contain study ingredients
  Interventions: Dietary Supplement: Dietary supplement liquid shot beverage products
- Experimental Product 1 (Experimental): Developmental liquid shot beverage product: prototype 60ml product that contains study ingredients
  Interventions: Dietary Supplement: Dietary supplement liquid shot beverage products
- Experimental Product 2 (Experimental): Developmental liquid shot beverage product: prototype 60ml product that contains study ingredients
  Interventions: Dietary Supplement: Dietary supplement liquid shot beverage products

INTERVENTIONS:
Dietary Supplement: Dietary supplement liquid shot beverage products — Participants will use their product as instructed for 3 of the 4 study weeks

SUMMARY:
A home placement, randomized, double blind, placebo-controlled, study to determine the effect of dietary liquid shot beverage products on self-reported measures of sleep, stress and mood on generally healthy participants with current self-reported mild/moderate sleep difficulties (but not clinical insomnia) and mild/moderate stress.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy participants, between 18 and 55 years of age.
* Participants who are not clinical insomniacs (as determined by a medical professional in the last 12 months, or who meets the ISQ criteria in screening).
* Participants who are in good self-reported physical and mental health.
* Participants with current self-reported mild/moderate sleep difficulties wishing to improve their sleep (as determined by an AIS score of 7 or more, but 14 or less).
* Participants with current self-reported mild/moderate stress wishing to improve their stress level (as determined by a PSQ raw score of 38 or higher).
* Participants that are willing to not use other new dietary supplements throughout the study but continue to use their normal dietary supplements (if any) as per their normal routine.
* Participants who can provide written informed consent to participate in the study and will have agreed to abide by the study restrictions, requirements and protocol.
* Participants must, in the opinion of the Principal Investigator (or designee), demonstrate the ability to comprehend the informed consent form (ICF), understand and comply with the requirements of the study, and be judged suitable for the study.
* Participants must be available to complete the study.
* Participants must be willing to abstain from alcohol after 6 pm each day.
* Participants must consume less than 400 mgs of caffeine per day.
* Participants must consume 7 servings or less of alcohol in a typical week

Exclusion Criteria:

* Participants that are not US citizens or residents.
* Participants that have a medical condition, including but not limited to heartbeat/rhythm irregularities, past heart attacks, been diagnosed with heart disease, seizure disorder, autoimmune disease, kidney disorder or impairment, chronic sinus condition, liver condition, blood clotting disorder, endocrine-related medical diagnosis (such as diabetes, thyroid, etc.), asthma/emphysema/COPD, serious health condition (i.e., cancer, etc.), blindness, insomnia, narcolepsy, anxiety, depression, hypertension, or deafness.
* Participants that have a BMI outside the range of 18.5 to 35.
* Participants that do not sleep during the night, do not work day-shift hours, or have other factors that impact their sleep schedule such as an inconsistent work schedule, or dealing with chronic pain or having a sleep disorder (such as Night Terrors, Narcolepsy, Insomnia, or Sleep Apnoea).
* Participants that do not have any difficulty sleeping.
* Participants that use recreational drugs or that are currently taking prescription medication (except for a contraceptive).
* Participants that are pregnant, breastfeeding (or pumping/expressing) or intend to become pregnant within the next six months.
* Participants that currently use cannabinoid products, smoke cigarettes or use any tobacco or nicotine products.
* Participants that are allergic or sensitive to any of the product ingredients.
* Participants that are currently or have participated in sleep-related studies or any product research studies in the last 30 days.
* Participants that currently work (or who have an immediate family member who works) for a market research, marketing, advertising, public relations, pharmaceutical, food/beverage or tobacco company.
* Participants that use sleep aids every night or multiple times a week.
* Participants who are unwilling or unable to comply with the study requirements and restrictions including those outlined in the Participant Handbook.
* Participants that are traveling over the next 4-6 weeks, to an extent where the time zone difference would impact their regular sleep schedule

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Sleep Disturbance | Time points: Week 1, 2, 3 and 4
  Change in Patient-Reported Outcomes Measurement Information Systems (PROMIS) - Sleep disturbance 8A
  Scores range from 8-40, where lower scores indicate lower sleep disturbance

SECONDARY OUTCOMES:
Sleep Impairment | Time points: Weeks 1, 2, 3, and 4
  Change in Patient-Reported Outcomes Measurement Information Systems (PROMIS) - Sleep-related impairment score 8A
  Scores range from 8-40, where lower scores indicate lower sleep impairment
Insomnia Severity Scores range from 0-24, where lower scores indicate lower insomnia severity | Time points: Weeks 1, 2, 3, and 4
  Change in Athens Insomnia Scale (AIS) score
  Scores range from 0-24, where lower scores indicate lower insomnia severity
Restorative Sleep Scores range from 0-100, where higher scores indicate better restorative sleep | Time points: Weeks 1, 2, 3, and 4
  Change in Restorative Sleep Questionnaire (RSQ) score
  Scores range from 0-100, where higher scores indicate better restorative sleep
Contentedness/Anxiety Scores range from 6-24, where lower scores indicate lower levels of state anxiety | Time points: Weeks 1, 2, 3, and 4
  Change in 6-item State Anxiety Inventory (STAI) - State Only portion
  Scores range from 6-24, where lower scores indicate lower state anxiety
Profile of Mood States (POMS 35 Item version) | Time points: Weeks 1, 2, 3, and 4
  Change in the following POMS scores:
  * Anger
  * Confusion
  * Depression
  * Fatigue
  * Tension
  * Vigor
  * Friendliness
  Scores range from 0-20 for each score
  • Total Mood Disturbance
  Scores for total mood disturbance range from -20 to 100
Daily Sleep diary | Time points: averages of weeks 1, 2, 3, and 4 (Sunday night - Thursday night consumption only, reported on Monday - Friday mornings)
  Change in the following:
  * Total sleep time the previous night (self-report estimated in 15 minute increments)
  * Satisfaction with how long it took to fall asleep the previous night (7-point likert scale, where higher scores indicate higher satisfaction with how long it took to fall asleep)
  * Time spent awake during the night (self-reported estimate in estimated minutes/hours)
  * Sleep quality VAS (scores range from 0-100, where higher scores indicate higher perceived sleep quality)
  * Relaxation upon waking VAS (scores range from 0-100, where higher scores indicate higher relaxation)
  * Refreshment upon waking VAS (scores range from 0-100, where higher scores indicate higher refreshment)
  * Alertness upon waking VAS (scores range from 0-100, where higher scores indicate higher alertness)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Niedziela, PhD, Principal Investigator — HCD Research
Locations (1):
- Sago Atlanta - The Palisades Complex, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided